CLINICAL TRIAL: NCT03900520
Title: Evaluating Pneumococcal Conjugate Vaccine (PCV) Impact on Pneumonia and Pneumococcal Carriage Outcomes in India in Children 1-35 Months in India: Pneumonia Research and Vaccine Impact League
Brief Title: Pneumonia Research and Vaccine Impact League
Acronym: PREVAIL
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Maulana Azad Medical College (Other); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 11740
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Pneumonia
Keywords: pneumococcal conjugate vaccine; vaccine impact; radiographic pneumonia; hospitalization; nasopharyngeal swab; India; cost of illness; pneumococcal carriage; pneumococcal serotypes; pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pneumonia group (PREVAIL-Pneumo): Children aged 1-35 months with pneumonia or lower respiratory tract infection hospitalized or recommended for hospitalization
- Community group (PREVAIL-Community): Children aged 1-35 years living in the community with no known systemic illness
- Economic group (PREVAIL-Econ): PREVAIL-Pneumo-enrolled children hospitalized for pneumonia

SUMMARY:
The leading cause of severe respiratory disease and death in young children is Streptococcus pneumoniae (pneumococcus). An estimated one-fifth of global childhood pneumococcal-related deaths occurred in India. The pneumococcal conjugate vaccine (PCV) is a primary prevention tool against pneumococcal disease that is safe and effective and has been in use in many countries. In alignment with the Government of India's rollout of PCV sub-nationally in selected districts and states, this two-year observational study will use a non-interventional, observational prospective study design to evaluate the impact of PCV in 7 sites in India (5 hospitals and 2 community sites) by assessing clinical and serotype-specific outcomes that include hospitalized pneumonia and community pneumococcal carriage. A sub-study to assess the cost of illness of pneumonia will also be conducted. This study is anticipated to provide data to support sustainability of PCV expansion and disease surveillance in India.

DETAILED DESCRIPTION:
Streptococcus pneumoniae (pneumococcus) is the leading cause of severe respiratory disease and death in young children, and is also responsible for other serious diseases such as meningitis and sepsis. Global disease burden models for the year 2015, estimate that 20 percent of global childhood pneumococcal deaths occurred in India. Data from India indicate that available pneumococcal conjugate vaccines (PCV) include serotypes that account for 66 to 74 percent of invasive pneumococcal disease (IPD) in young children. The 2017 PCV launch into the national immunization schedule in selected high-burden states was poised to successfully combat the pneumococcal disease burden in the country once scale-up of vaccine coverage takes place. The Government of India has recommended robust evaluation of PCV impact to facilitate national rollout and sustained use of PCV.

This study aims to evaluate the impact of PCV introduction to the national immunization program. The investigators propose to quantify the impact of PCV on pneumonia and other acute respiratory infections resulting in hospitalization and on community carriage of pneumococci. Hereafter, in reference to the proposed study, the investigators use the term 'pneumonia' to denote to a group of physician-based diagnoses representing a range of acute respiratory illness including pneumonia. Specifically, the investigators propose to measure differences in the proportion of pneumonia hospitalizations in children 1-35 months colonized with vaccine-serotype (VT) pneumococcus, as well as differences in VT pneumococcal nasopharyngeal (NP) colonization in the community, comparing children enrolled at sites where PCV has been introduced (PCV sites) to children at sites where PCV has not yet been introduced (non-PCV sites). The health economic aims will consist of assessing the cost of illness of pneumococcal disease, and economic cost of pneumococcal disease and pneumonia hospitalization. The investigators have designed this portfolio of PCV impact evaluations within the context of PCV introduction and rollout in six selected states in India, mindful of the need for baseline data, the staggered plan for PCV roll-out, variance of cost-generating events, and the inherent biases of non-interventional studies with outcomes that are not specific for pneumococcal disease and that may be subject to secular trends and possible confounders. The study sites are located in New Delhi and within three of the six states that were included in the PCV rollout plan starting in 2017. The investigators plan this as a two-year study that will include data from both PCV sites and non-PCV sites, the comparison of which will allow an assessment of vaccine impact. Active study sites will be located in Delhi; Agra in Uttar Pradesh state (non-PCV-using); Bhopal in Madhya Pradesh state; and Jaipur in Rajasthan state (PCV-using). Community enrollment will take place in two demographic survey sites in Bhopal and Delhi, and economic assessment will take place in four hospital sites. Sites will use a common protocol to identify and recruit children, obtain nasopharyngeal swabs for colonization studies, and run validated laboratory tests. A reference laboratory will provide pneumococcal serotyping results, nasopharyngeal quantification of pneumococcus, and provide site laboratory oversight.

These data will provide evidence to policy makers on changes in pneumococcal disease burden in young children, pneumococcal community transmission changes as a result of PCV introduction, that can help policy makers support, optimize, and advocate for the expansion of the PCV immunization program in India and in other countries.

The primary objectives of PREVAIL are as follows:

1. Quantify the difference in the proportion of hospitalized pneumonia cases 1-35 months of age carrying a vaccine-type pneumococcus in the nasopharynx in cases enrolled at sites that have introduced PCV into the national immunization program compared to cases enrolled at sites that have not introduced PCV
2. Quantify the difference in the proportion of children in the community 1-35 months who are colonized with vaccine-type pneumococcus enrolled at a site that has introduced PCV into the national immunization program compared to the proportion of children colonized with vaccine-type pneumococcus enrolled at a site that has not introduced PCV
3. Determine the overall economic impact of PCV by: (i) Estimating the total cost of hospitalized pneumonia in children 1-35 months from the healthcare system and household perspectives; and (ii) Estimating the proportion of households facing catastrophic health spending and medical impoverishment from out-of-pocket health expenses due to hospitalized pneumonia in children 1-35 months.

Secondary objectives are evaluated within each of the four groups, and are;

1. Assess the difference in mortality and occurrence of illnesses within 3 months of hospital discharge among children aged 1-35 months presenting with pneumonia in PCV-using sites compared to children at non-PCV sites.
2. Quantify the difference in proportion among hospitalized cases aged 1-35 months with alveolar consolidation detected on radiography in PCV-using sites compared to children at non-PCV sites.
3. Quantify the difference in proportion among hospitalized cases aged 1-35 months with hypoxemia (oxygen saturation<90%) in PCV-using sites compared to children at non-PCV sites.
4. Quantify the difference in proportion of hospitalized cases aged 1-35 months that are vaccinated at PCV-using sites (indirect cohort method to assess vaccine effectiveness) between the following groups:

   1. Carrying a VT vs. carrying a non-VT serotype
   2. With vs. without alveolar consolidation
   3. With vs. without hypoxemia

ELIGIBILITY:
PREVAIL-Pneumo:

Inclusion criteria:

* Age 1-35 months
* Admitting diagnosis is pneumonia or lower respiratory tract illness/infection Written informed consent obtained from parent or legally authorized representative

Exclusion criteria:

* Discharged as an PREVAIL case in the last 90 days

PREVAIL-Community:

Inclusion criteria:

* Age 1-35 months with no systemic illness (mild respiratory illness is not an exclusion criteria)
* Written informed consent obtained from parent or legally authorized representative

Exclusion criteria:

* Known underlying serious disease (e.g., congenital heart diseases, immunodeficiency disorders, sickle cell anemia etc.) which may negatively influence the participant's ability to participate in the study

PREVAIL-Econ:

Inclusion criteria:

* Currently enrolled into the PREVAIL study

Ages: 1 Month to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: There are three cohorts/groups that are recruited:
  PREVAIL-Pneumo: Cases aged 1-35 months of age hospitalized with physician-diagnosed pneumonia or lower respiratory tract infection.
  PREVAIL-Community: Children 1-35 months of age residing in the community with no systemic illness and randomly selected for inclusion into this group
  PREVAIL-Econ: A subset of cases enrolled into the PREVAIL-Pneumo study
Sampling Method: Probability Sample
Enrollment: 6004 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Pneumonia colonized by vaccine-type Streptococcus pneumoniae | 2 years (2 year period mentioned refers to the duration of the proposed study in total)
  PREVAIL-Pneumo: Proportion of children with physician-diagnosed pneumonia that are colonized in the nasopharynx with 'vaccine-type' pneumococcus among sites where PCV has been introduced compared to sites where PCV has not been introduced (includes 13 serotypes included in the 13-valent pneumococcal conjugate vaccine)
Community carriage of vaccine-type Streptococcus pneumoniae | 2 years (2 year period mentioned refers to the duration of the proposed study in total)
  PREVAIL-Community: Proportion of community children that are colonized in the nasopharynx with 'vaccine-type' pneumococcus enrolled at a site that has introduced PCV into the NIP compared to children enrolled at a site that has not introduced PCV (includes 13 serotypes included in the 13-valent pneumococcal conjugate vaccine)
Pneumonia and IPD cost of illness | 1 years (1 year period mentioned refers to the duration of the proposed study in total)
  PREVAIL-Econ: Determine the overall economic impact of PCV, including direct and indirect costs, both during hospitalization and longer-term expenditures at 3 months post hospitalization

SECONDARY OUTCOMES:
Pneumonia-Related Occurance of Illness | 2 years (2 year period mentioned refers to the duration of the proposed study in total)
  Difference in occurrence of illnesses within 3 months of hospital discharge among children 1-35 months presenting with pneumonia at sites that have introduced PCV into the national immunization schedule versus cases enrolled at sites that have not introduced PCV. (3 months refers to the duration each patient would be followed up for following discharge from the hospital)
Pneumonia-Related Mortality | 2 years (2 year period mentioned refers to the duration of the proposed study in total)
  Difference in mortality within 3 months of hospital discharge among children 1-35 months presenting with pneumonia at sites that have introduced PCV into the national immunization schedule versus cases enrolled at sites that have not introduced PCV. (3 months refers to the duration each patient would be followed up for following discharge from the hospital)
Radiographic pneumonia | 2 years (2 year period mentioned refers to the duration of the proposed study in total)
  Proportion of children with primary-end point pneumonia detected on radiography, at sites that have introduced PCV into the national immunization schedule versus cases enrolled at sites that have not introduced PCV.
Hypoxic Pneumonia | 2 years (2 year period mentioned refers to the duration of the proposed study in total)
  Proportion of children with hypoxemic (oxygen saturation<90 percent) among hospitalized pneumonia cases 1-35 months at sites that have introduced PCV versus cases enrolled at sites that have not introduced PCV.
Vaccine Effectiveness | 2 years (2 year period mentioned refers to the duration of the proposed study in total)
  Proportion of hospitalized cases 1-35 months that are vaccinated in PCV-using sites (indirect cohort method to assess vaccine effectiveness) between the following groups: (1) Carrying a VT vs. carrying a non-VT serotype, (2) With vs. without alveolar consolidation, (3) With vs. without hypoxemia.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Shet, MD, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Maulana Azad Medical College, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided